CLINICAL TRIAL: NCT02809963
Title: A Randomized, Double-blind, Placebo-controlled Study of the Effect of Mineralocorticoid Receptor Antagonists in Type 2 Diabetes Patients on Myocardial Function, Glucose and Fat Metabolism (The MIRAD-study)
Brief Title: Mineralocorticoid Receptor Antagonists in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Marie Louise Johansen, MD, PhD student, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-002519-14
Record Dates: First submitted 2016-06-16; First posted 2016-06-22 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eplerenone (Active Comparator): Eplerenone 50 mg tablets. 2-4 tablets once daily for 26 weeks
  Interventions: Drug: Eplerenone
- placebo (Placebo Comparator): sugar pill manufactured to mimic Eplerenone 50 mg tablet. 2-4 tablets once daily for 26 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eplerenone — 50 mg tablets, oral use.
  Arms: Eplerenone
Drug: Placebo — 50 mg tablets, oral use
  Arms: placebo

SUMMARY:
The aim of this study is to investigate the effect of selective blocking of the mineralocorticoid receptor in patients with type 2 diabetes on insulin resistance, lipid metabolism and myocardial function.

DETAILED DESCRIPTION:
In this randomized, double-blind, placebo-controlled study we want to investigate the effect of mineralocorticoid receptor antagonists in type 2 diabetes patients on myocardial function, glucose and fat metabolism.

Background The mortality rate in T2 DM is still increased by almost a factor 2 although poly pharmacological therapy of risk factors has been recommended for years. Treatment with MR antagonists in patients with primary hyperaldosteronism and systolic heart failure improves insulin resistance, myocardial function and prognosis. Further, recent evidence has suggested that aldosterone participates in the regulation of glucose and lipid metabolism, as MR expression has been identified in adipocytes and beneficial metabolic effects of selective MR blockade has been demonstrated in several animal models. Notably, there is no available data in humans with T2DM.

A key feature of T2 DM is altered body composition characterized by increased metabolic active visceral adipose tissue (VAT) and increased fat content of the liver, which has been associated with cardiac dysfunction and outcome. Gold standard for measurement of VAT is magnetic resonance imaging (MRI), and proton MRI spectroscopy can quantitatively measure fat content in the liver with high precision. The pathogenesis of myocardial dysfunction in T2DM is linked with insulin resistance (IR) of adipose tissue mediating increased supply of free fatty acids and intra myocardial lipid accumulation. Thus, beneficial effects of lipid metabolism could in theory indirectly improve myocardial function in type 2 diabetics.

Global longitudinal strain (GLS) is a validated method for evaluating regional and global function of the left ventricle, which is a strong predictor of incident HF in patients with myocardial infarction and closely related with plasma NT-proBNP concentrations.

Hypothesis Selective blocking of the MR receptor in patients with T2 DM improves insulin resistance, lipid metabolism and myocardial function.

Objectives To investigate the effect of Eplerenone 100-200 mg once daily compared to placebo in patients with type 2 diabetes with regard to glucose and lipid metabolism, myocardial function and structure, and vascular function.

The primary objective is to investigate the effect of Eplerenone 100-200 mg once daily compared to placebo on changes in liver fat content.

Design A single center, randomized, double blinded placebo controlled trial. Patients with T2 DM and high risk of cardiovascular disease will be randomized to either Eplerenone 100-200 mg or placebo daily for 26 weeks. Patients will be investigated at baseline and after 26 weeks.

A total of 130 patients with type 2 diabetes will be included.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the written patient information and to give informed consent
* Type 2 diabetes mellitus (WHO criteria), diagnosed at least 3 months prior to baseline
* Blood pressure treatment according to standard guidelines
* Negative pregnancy test (fertile women)
* Be willing to change/pause potassium sparing medication
* Age 18-85 years
* Patients must have high cardiovascular risk factors, defined as one of the following:

NT-proBNP ≥ 70 pg/ml (taken within the last 6 months prior to baseline) Albuminuria ( albumin/creatinine ratio ≥ 30 mg/g Confirmed history of myocardial infarction (≥ 3 months prior to baseline) Or patient discharged from hospital with a documented diagnosis of unstable angina within 24 months prior to baseline Evidence of coronary artery disease by CAG in 1 or more major coronary arteries OR at least one of the following: a positive noninvasive stress test, OR a positive stress echocardiography showing regional systolic wall motion abnormalities, OR a positive scintigraphy test showing stress-induced ischemia History of ischemic or hemorrhagic stroke (≥ 3 months prior to informed consent) Presence of peripheral artery disease (symptomatic or not ) documented by either: previous limb angioplasty, stenting or bypass surgery; or previous limb or foot amputation due to circulatory insufficiency; or angiographic evidence of significant (≥ 50%) peripheral artery stenosis in at least one limb; or evidence from a non-invasive measurement of significant (≥50% or as reported as hemodynamically significant) peripheral artery stenosis in at least one limb; or ankle brachial index of ≤ 0.9

Left ventricle hypertrophy:

Documented at echocardiography ECG: R-spike in V5/V6 ≥ 25 mm or S-spike in V1 + R-spike in V5/V6 ≥ 35 mm Patients both with and without a cardiovascular risk factor can be randomized to the fat biopsy sub study.

Exclusion Criteria:

* Allergic to the study medication
* Systolic HF (LVEF ≤ 40%)
* Impaired kidney function, eGFR ≤ 40 ml/min
* Severe liver insufficiency (Child-Pugh class C)
* Treatment with MR antagonist within 3 months prior to baseline
* Treatment with both ACE inhibitors and Angiotensin II Receptor blockers.
* Serum-potassium ≥ 5.0 mmol/l
* Serum-sodium ≤ 135 mmol/l
* Myocardial infarction, unstable angina pectoris or bypass graft surgery within 3 months prior to baseline
* Persistant atrial fibrillation (except for the fat biopsy sub population)
* ECG showing malign ventricular arrhythmia or prolonged QT-interval (> 500ms)
* Untreated heart valve disease
* ICD-unit/pacemaker
* Pregnancy or desire hereof or breastfeeding
* Women in the fertile age not using safe contraceptives (spiral, hormonal contraceptives)
* Cancer unless complete remission ≥ 5 year
* Alcohol-/drug-abuse
* Inflammatory bowel disease
* Other concomitant disease or treatment that according to the investigator's assessment makes the patient unsuitable to participate in the study
* Simultaneous participation in another clinical study
* Treatment with CYP3A4-inhibitors (e.g. itraconazol, etoconazol, ritonavir, nelfinavir, clarithromycin, telithromycin and nefazodon)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-11; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Liver fat content | 26 weeks
  changes in liver fat content by proton MR spectroscopy

SECONDARY OUTCOMES:
Fat mass distribution | 26 weeks
  Changes in body fat distribution (total body fat, visceral fat, subcutaneous fat)
insulin resistance | 26 weeks
  Changes in insulin resistance by HOMA and Matsuda index
Urinary albumin/creatinine ratio | 26 weeks
  changes in Urinary albumin/creatinine ratio
Biomarkers of adipocyte function | 26 weeks
  Changes in biomarkers of adipocyte function (adiponectin, leptin, FGF-21, TNF-alfa, FFA, IL-6, MCP-1, MAC-1)
24 Hour blood pressure | 26 weeks
  changes in 24 Hour blood pressure
Global longitudinal strain (GLS) | 26 weeks
  changes in global longitudinal strain by echocardiography
systolic and diastolic function og left ventricule | 26 weeks
  changes in systolic and diastolic function of left ventricule by echocardiography
Regional and global fibrosis by cardiac magnetic resonance | 26 weeks
  changes in regional and global fibrosis using Late gadolineum enhancement cardiac magnetic resonance
biomarkers of myocardial stress and fibrosis | 26 weeks
  changes in biomarkers of myocardial stress and fibrosis (NT-proBNP, MR-proANP, galectin-3, GDF-15, MR-proADM)
pulse wave analysis | 26 weeks
  changes in pulse wave analysis
Quality of life | 26 weeks
  changes in quality of life using WHO-5
Diabetes related changes in quality of life | 26 weeks
  changes in quality of life using W-BQ12
kidney function | 26 weeks
  changes in creatinine and eGFR
potassium | 26 weeks
  changes in potassium

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev and Gentofte Hospital, Department of Endocrinology and Metabolism, Department of internal medicine,, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No